CLINICAL TRIAL: NCT06567587
Title: Assessing the Efficacy of Dexmedetomidine in Alleviating Agitation for Exacerbated COPD Patients Who Are Treated for Psychosis Requiring Non- Invasive Ventilation
Brief Title: Dexmedtomodine Effect on Agitated Psychotic Patients Suffer COPD
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Collaborators: Laila Ahmed Abd-Elmotaleb El-Ahwal (Unknown); Marwa Ahmed Abogabal (Unknown)
Responsible Party: Principal Investigator, Mohamed Zakarea Wfa, Lecturer of Anesthesia, Surgical ICU and Pain Medicine, Tanta University
Other Study IDs: 36264PR678/5/24
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Response of Agitated Patients to Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Group I: 35 Patients came to ICU with exaggerated COPD and suffer delirium and agitation
  Interventions: Drug: Dexmedetomidine; Device: BIPAP
- Group II: 35 psychotic patients on medical treatment came to ICU with exaggerated COPD and suffer delirium and agitation.
  Interventions: Drug: Dexmedetomidine; Device: BIPAP

INTERVENTIONS:
Drug: Dexmedetomidine — Effect o dexmedetomine on agitated normal and psychotic patients on BIPAP who are suffer exaggerated COPD
  Other Names: Precedex
Device: BIPAP — Put exaggerated COPD patients on non invasive ventillation
  Other Names: Non invasive ventiillation

SUMMARY:
Many studies approved dexmedetomodine as a drug controlled agitation for psychotic patients and also for patients on non invasive ventilation.

So we study the same effect on agitated patients who are on non invasive ventilation and also suffer of psychosis as agitation become more aggressive than usual

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) characterized by progressive airflow limitation and tissue destruction as there are structural lung changes due to chronic inflammation from prolonged exposure to noxious particles or gases most commonly cigarette smoke. Chronic inflammation causes airway narrowing and decreased lung recoil. The disease often presents with symptoms of cough, dyspnea, and sputum production and may be exacerbated to cause respiratory failure. Acute exacerbations of chronic obstructive pulmonary disease can range from self-limited diseases to episodes of florid hypercapnic respiratory failure requiring non-invasive ventilation and late may be mixed type of respiratory failure due to hypercarbia and hypoxia and patients may need invasive ventilation.Hypercapnia generates increased sympathetic tone and decreased parasympathetic tone, it may be due to increases in brain glutamine and gamma-aminobutyric acid and this causes state of agitation and delirium. agitated COPD patients present a unique challenge due to the interplay between respiratory distress and psychiatric symptoms, which can complicate treatment.

Dexmedetomidine, a selective alpha-2 adrenergic agonist with sedative and analgesic properties by decreasing glutamate release and also it lacks GABA receptor modulation or cholinergic receptor activity. Additionally, dexmedetomidine may promote natural sleep patterns through stimulation of α 2 receptors leading to inhibition of noradrenergic neurons in the locus ceruleus and disinhibition of GABA neurons in the ventrolateral preoptic nucleus.The RASS is a 10-point scale ranging from -5 to +4. Levels -1 to -5 denote 5 levels of sedation, starting with"awakens to voice" and ending with "unarousable. Levels +1 to +4 describe increasing levels of agitation.

The lowest level of agitation starts with apprehension and anxiety, and peaks at combative and violent. RASS level 0 is "alert and calm. Psychiatric disorders are a category of behavioral and psychological syndromes that reflect underlying psychobiological dysfunction, leading to significant distress and impairment . Patients with pre-existing psychiatric disorders have an increased risk of poor health outcomes during an ICU stay, including increased odds of mechanical ventilation, organ dysfunction, and mortality, compared to patients without psychiatric disorders .This study aims to fill this gap by assessing the impact of dexmedetomidine on both respiratory parameters and psychiatric symptoms, with the goal of improving overall patient outcomes and guiding future treatment approaches in this complex.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 60 years, ASA III (agitated and exacerbated COPD patients).

Exclusion Criteria:

* Patients with GCS < 8 (need invasive ventilation).

  * Failure of non-invasive ventilation.
  * Patients with fascial trauma or surgery.
  * Patients with esophageal varices.
  * Patients with recent GIT surgeries.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who will meet the previous criteria will be enrolled in the study. Patients will be classified into two equal groups; 35 patients will be enrolled in each group; all patients will receive loading dose of dexmedetomidine 1 μg/kg in 10 min then maintenance dose 0.2-0.7 μg/kg/hr till obtain adequate sedation level guided by Richmond agitation score.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 6 months
  failure rate of patients necessitates invasive ventilation after non-invasive ventilation.

SECONDARY OUTCOMES:
Secondary outcome | 6 months
  Richmond agitation score.
  • Effective doses of dexmedetomidine are needed to control agitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Dexmedetomidine effect on agitated psychotic COPD patients on non invasive ventillation